CLINICAL TRIAL: NCT01772966
Title: Generalizing a Valid Control Manipulation to a Multiple Operator, Longitudinal Randomized Controlled Study for Chronic Neck Pain
Brief Title: Chiropractic Manual Therapy and Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122008; R01AT007311-01 (NIH)
Record Dates: First submitted 2012-09-21; First posted 2013-01-21 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: neck; pain; chronic; manipulation; control; randomized trial
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal manipulation (Experimental): Participants will receive spinal manipulation delivered as segmental thrust to a specific site in the neck. They will receive three intervention sessions over 7-10 days.
  Interventions: Procedure: Spinal manipulation
- Control manipulation (Sham Comparator): Participants will receive spinal manipulation delivered as non-segmental thrust to the neck. They will receive three intervention sessions over 7-10 days.
  Interventions: Procedure: Spinal manipulation

INTERVENTIONS:
Procedure: Spinal manipulation

SUMMARY:
Eligible subjects with chronic neck pain will be randomly allocated to one of two intervention groups: real vs control spinal manipulation. They will receive three intervention sessions.

H1: Chronic neck pain patients treated longitudinally over a series of three encounters in one week by random assignment to treatment group with either of the dual delivery procedures (Intervention 1=typical-control or Intervention 2=control-control) will have a 50% error rate of self-report of group allocation at exit interview.

H2: Patients treated by the typical-control dual procedure over a typical sequence of encounters (3 times in one week) will show statistically significant improvement in clinical outcomes; defined quantitatively by visual analogue pain scale (VAS), Neck Disability Index (NDI), range of motion and pressure algometry; compared to those treated by the control-control dual procedure.

H3: Patients stratified by 'a priori' patient expectation for treatment outcome will show no significant difference in self-report of group allocation or clinical outcome measures.

A total of 372 subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 21 to 60 years of age
* Chronic neck pain
* Neck pain duration greater than 6 weeks
* Numeric Rating Scale greater than 30, less than 65
* Pain distribution between nuchal ridge and spine of the scapula
* Pain aggravated by local provocation maneuvers at single motion segment
* Antero-posterior glide
* Paraspinal tenderness
* Negative provocative maneuvers at adjacent segment
* Able to tolerate neck movement to 50 percent normal in all directions

Exclusion Criteria:

* Worker's compensation or other medico-legal claim
* Cervical spine surgery or fracture or dislocation
* Uncontrolled hypertension (Blood Pressure over 140 over 90)
* Stroke or Transient Ischemic Attack
* Upper respiratory infection within 4 weeks
* Severe degenerative disease of the cervical spine
* New or significantly altered pattern of headache complaint
* Connective tissue disease
* Primary fibromyalgia
* Metabolic or metaplastic bone disease
* Whiplash injury within 12 months
* High cholesterol levels not well-managed medically
* Cardiovascular surgery in the past 6 months or planned
* Use of narcotic analgesic, prescription anti-inflammatory, or muscle relaxants, anti-convulsants
* Angina pectoris
* Dizziness
* Tinnitus
* Blurred vision, vertigo, undiagnosed sensory and motor disturbances
* Radicular symptoms and signs
* Current use of anticoagulant therapy
* Upper respiratory infection
* Neck pain on provocation greater than 7 out of 10
* Provocation of radicular pain or sensory disturbance
* Hypermobility of multiple peripheral joints,
* Physical or mental impairment precluding following instructions or participating -in supine recumbent postures

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2013-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Group registration | At exit assessment following the third intervention session
  Participants will be asked to identify which of the two interventions they feel they received.

SECONDARY OUTCOMES:
Pain severity | 1. at baseline, and 2. At exit assessment following the third intervention session
  Pain scores on the PROMIS pain severity instrument.
Improvement | At exit assessment following the third intervention session
  Participants will be asked to rate their level of improvement on the The Global Rating of Change instrument.
Disability | 1. at baseline, and 2. At exit assessment following the third intervention session
  Participants will score the The Neck Disability Index (score out of 50).
Tenderness | 1. at baseline, and 2. At exit assessment following the third intervention session
  Pressure algometry over a single specified spinal site will be used to measure tenderness in kg/sq.sm.

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | Daily over 7-10 days.
  All adverse events will be described and tallied. Adverse events will be categorized in two modes: 1] Serious vs. Not Serious, and, 2] Attributable to the trial vs. Not Attributable. Both the absolute number of adverse events as well as the percentage of subjects experiencing an adverse event will be reported.
Expectations related to improvement | Baseline
  Participants' expectations of the efficacy of the interventions will be obtained at baseline with the protocol of Fulda et al.

CONTACTS AND LOCATIONS:
Overall Officials: Howard T Vernon, DC, PhD, Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada

REFERENCES:
- [Result] Vernon H, MacAdam K, Marshall V, Pion M, Sadowska M. Validation of a sham manipulative procedure for the cervical spine for use in clinical trials. J Manipulative Physiol Ther. 2005 Nov-Dec;28(9):662-6. doi: 10.1016/j.jmpt.2005.07.020. PMID 16326235